CLINICAL TRIAL: NCT02950064
Title: Escalation Study of BTP-114 in Patients With Advanced Solid Tumors and BRCA or DNA Repair Mutation
Brief Title: A Study to Determine the Safety of BTP-114 for Treatment in Patients With Advanced Solid Tumors With BRCA Mutations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Placon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-114-001
Record Dates: First submitted 2016-10-05; First posted 2016-10-31 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms
Keywords: BRCA; BRCA1; BRCA2; Pancreatic cancer; Ovarian cancer; Castrate resistant prostate cancer; Triple negative breast cancer; Breast cancer; DNA repair mutation-positive solid tumors
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTP-114 (Experimental): Intravenous (IV) treatment n 21-day cycles
  Interventions: Drug: BTP-114

INTERVENTIONS:
Drug: BTP-114 — Part 1 (Escalation) IV treatment of BTP-114 in 21-day cycles. Doses will be increased in sequential cohorts until the maximum tolerated dose is determined which will lead to the recommended phase 2 dose
  Part 2 (Expansion) 5 cohorts of patients will be treated at the RP2D of IV BTP-114 in 21-day cycles for the tumor types pancreatic cancer, castration-resistant prostate cancer, ovarian cancer, triple-negative breast cancer and deoxyribonucleic acid (DNA) repair mutation-positive advanced solid tumors.

SUMMARY:
This is a phase 1, Open-label, multicenter Dose Escalation study of BTP-114, a novel platinum product, in patients with advanced solid tumors and BRCA or other DNA repair mutation. This clinical study is comprised of 2 sequential parts: Part 1 (Dose Escalation) and Part 2 (Expansion). The purpose of this study is to evaluate the safety, pharmacokinetics and the anti-cancer activity of BTP-114.

ELIGIBILITY:
INCLUSION:

All Patients

1. Male or female aged ≥18 years.
2. ECOG PS score of 0-1.
3. Adequate organ function.
4. Ability to understand and willingness to sign informed consent form prior to initiation of study procedures.
5. Measurable disease per RECIST, OR for patients with a primary diagnosis of castration resistant prostate cancer, progressive disease (PD) by prostate surface antigen (PSA) or imaging in the setting of medical or surgical castration.
6. Documented BRCA mutation, with the following exceptions: a) Patient is intended to be enrolled in a Single-patient Cohort; b) Patient has an advanced DNA repair mutation-positive solid tumor and is intended to be enrolled in Expansion Cohort 5.

   Patients in the Dose-escalation Phase:
7. Locally advanced solid tumor other than a primary central nervous system (CNS) tumor for which the patient has received ≤3 prior lines
8. Confirmed solid tumor in one of the following categories:

   * BRCA mutation-positive pancreatic cancer for which the patient received up to 1 prior line of cytotoxic chemotherapy in the advanced disease setting.
   * Advanced BRCA mutation-positive castration-resistant prostate cancer (CRPC) for which the patient received up to 2 prior lines of cytotoxic chemotherapy in the advanced disease setting.
   * Advanced BRCA mutation-positive ovarian cancer for which the patient received up to 3 prior lines of cytotoxic chemotherapy in the advanced disease setting.
   * Advanced BRCA mutation-positive triple-negative breast cancer (TNBC) for which the patient received up to 3 prior lines of cytotoxic chemotherapy in the advanced disease setting.
   * Advanced DNA repair mutation-positive solid tumors, including, but not limited to BRCA and non-BRCA DNA mutations, who have received up to 3 prior lines of cytotoxic chemotherapy in the advanced disease setting. DNA-repair mutations may include, but are not limited to ATM, CHEK2, PALB2, and RAD51D. Abnormal homologous repair deficiency (HRD) tests will also be allowed.

Note that in both dose escalation and dose expansion portions of the study, prior targeted therapy including prior poly ADP ribose polymerase (PARP) inhibitor therapy, prior immunotherapy, or prior hormonal therapy is permissible. Patients with castration resistant prostate cancer may have received unlimited prior hormonal therapies.

EXCLUSION:

1. History of leptomeningeal disease or spinal cord compression.
2. Underwent major surgery within 4 weeks before first treatment.
3. Received cancer-directed therapy 14 days (6 weeks for mitomycin C and nitrosoureas) before start of treatment.
4. Grade 2 or greater peripheral neuropathy at start of treatment.
5. If female, pregnant or breast-feeding.
6. Known human immunodeficiency virus (HIV) infection or hepatitis B or C infection
7. Any primary brain tumor (e.g., astrocytoma, glioblastoma).
8. Hypersensitivity or history of anaphylactic reaction to any platinum-containing agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Maximum tolerated dose (MTD) of BTP-114 determined during the dose escalation phase of study based on number of patients experiencing a dose-limiting toxicity. | From the date of the first dose up to approximately 52 weeks.
Part 1 - Recommended Phase 2 Dose (RP2D) of BTP-114 based on the MTD, review of adverse event data and review of AUC, Tmax and t1/2 obtained from PK data during the dose escalation phase of the study. | From the date of the first dose up to approximately 52 weeks.
Part 1 - Number of patients experiencing treatment-related adverse events as assessed by CTCAE v4.3 during the study. | From the date of first dose up to approximately 52 weeks.
Part 2 - Proportion of patients with an objective response (ORR) using the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 or the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria. | From the date of the first dose to documented disease progression assessed up to approximately 52 weeks.
Part 2 - Proportion of patients whose disease is controlled (DCR) using RECIST, Version 1.1 or PCWG2 criteria. | From the date of the first dose to documented disease progression assessed up to approximately 52 weeks.
Part 2 - Duration of response (DOR) measured from the date of first CR or PR until the first date of progressive disease or death from any cause. | Assessed up to approximately 52 weeks.
Part 2 - Progression-free survival (PFS) measured as the time from the date of initiation of BTP-114 treatment to the documented disease progression (PD) or death from any cause. | Assessed up to approximately 52 weeks.

OTHER OUTCOMES:
Part 1 - Proportion of patients with an objective response (ORR) using the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 or the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria. | From the date of the first dose to documented disease progression assessed up to approximately 52 weeks.
Part 1 - Proportion of patients whose disease is controlled (DCR) using RECIST, Version 1.1 or PCWG2 criteria. | From the date of the first dose to documented disease progression assessed up to approximately 52 weeks.
Part 1 - Duration of response (DOR) measured from the date of first CR or PR until the first date of progressive disease or death from any cause. | Assessed up to approximately 52 weeks.
Part 1 - Progression-free survival (PFS) measured as the time from the date of initiation of BTP-114 treatment to the documented disease progression (PD) or death from any cause. | Assessed up to approximately 52 weeks.
Part 1 - Plasma Pharmacokinetics (PK) estimates of platinum concentration, Area under plasma Concentration (AUC) 0 to t. | Time points on Day 1, Day 3 or Day 4, Day 15 of Cycle 1 and Day 1 of subsequent cycles.
Part 1 - Plasma Pharmacokinetics (PK) estimates of platinum concentration, time of Maximum concentration (Tmax). | Time points on Day 1, Day 3 or Day 4, Day 15 of Cycle 1 and Day 1 of subsequent cycles.
Part 1 - Plasma Pharmacokinetics (PK) estimates of platinum concentration Half-life (T1/2). | Time points on Day 1, Day 3 or Day 4, Day 15 of Cycle 1 and Day 1 of subsequent cycles

CONTACTS AND LOCATIONS:
Overall Officials: Erika P Hamilton, MD, Principal Investigator — Tennessee Oncology
Locations (7):
- United States (7):
  - Placon Therapeutics Clinical Trial Site, Sarasota, Florida
  - Placon Therapeutics Clinical Trial Site, Boston, Massachusetts
  - Placon Therapeutics Clinical Trial Site, St Louis, Missouri
  - Placon Therapeutics Clinical Trial Site, Cleveland, Ohio
  - Placon Therapeutics Clinical Trial Site, Oklahoma City, Oklahoma
  - Placon Therapeutics Clinical Trial Site, Nashville, Tennessee
  - Placon Therapeutics Clinical Trial Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided